CLINICAL TRIAL: NCT01578369
Title: Pelvic Floor Muscle Training Included in General Fitness Classes is Effective in Primary Prevention of Urinary Incontince in Pregnancy. A Randomized Controlled Trial
Brief Title: Effect of Pelvic Floor Muscle Training Included in General Fitness Classes During Pregnacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Mireia Pelaez Puente, PhD, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 240/09B
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Pregnancy; Urinary Incontinence
Keywords: Urinary incontinence; Pregnancy; Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): Supervised exercise classes which included pelvic floor muscle training. 3 sessions per week. 55-60 min per session, with 10 minutes of pelvic floor muscle training. At least during 22 weeks.
  Interventions: Other: Exercise classes with pelvic floor muscle training
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Exercise classes with pelvic floor muscle training — Supervised exercise classes which included pelvic floor muscle training. 3 sessions per week. 55-60 min per session, with 10 minutes of pelvic floor muscle training. At least during 22 weeks.
  Arms: Exercise group

SUMMARY:
To investigate the effect of pelvic floor muscle training taught in a general exercise class during pregnancy to prevent urinary incontinence in nulliparous continent pregnant women.

DETAILED DESCRIPTION:
Pregnancy and childbirth are known risk factors for development of female urinary incontinence (UI). Studies have found that Pelvic Floor Mucle Trainig (PFMT) is effective in preventing and reducing UI during pregnancy and after childbirth. However, in a recent study, no effect was found when PFMT were taught in a general fitness class without former palpation of the pelvic floor muscles (Bo y Haakstad, 2011).

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous with singleton baby
* Not suffering from urinary incontinence
* Giving birth at Hospital Universitario de Fuenlabrada
* Able to comunicate in Spanish
* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines

Exclusion Criteria:

* Multiparity
* At risk of Premature birth
* Following another exercise program

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 169 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ICIQ-Urinary Incontinence Short Form Questionnaire | Week 10-14 gestation (baseline), week 36-39 (after intervention)

SECONDARY OUTCOMES:
Change from baseline in King's Health Questionnaire | week 10-14 of gestation (baseline), week 36-39 (after intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Universidad Politecnica de Madrid; Mireia Peláez, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Pelaez M, Gonzalez-Cerron S, Montejo R, Barakat R. Pelvic floor muscle training included in a pregnancy exercise program is effective in primary prevention of urinary incontinence: a randomized controlled trial. Neurourol Urodyn. 2014 Jan;33(1):67-71. doi: 10.1002/nau.22381. Epub 2013 Feb 6. PMID 23389863